CLINICAL TRIAL: NCT05184101
Title: INHALEd Nebulised Unfractionated HEParin for the Treatment of Hospitalised Patients With COVID-19 (INHALE-HEP) Australia
Brief Title: Inhaled Heparin for Hospitalised Patients With Coronavirus Disease 2019 (COVID-19)
Acronym: INHALE-HEP
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: COVID-19 hospitalisations limited in Australia, unable to recruit patients due to low numbers of hospitalisations.
Sponsor: Australian National University (Other)
Collaborators: The George Institute (Other); St George Hospital, Australia (Other); St Vincent's Hospital Melbourne (Other); John Hunter Hospital (Other Government); Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Frank van Haren, Professor, Australian National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INHALE-HEP Australia Version 3
Record Dates: First submitted 2022-01-06; First posted 2022-01-11 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: investigator-initiated, multi-centre, randomised, open-label trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulised heparin (Experimental): Participants assigned to 'nebulised heparin' will receive nebulised heparin in addition to the standard care required as determined by the treating team.
  Interventions: Drug: Unfractionated Heparin
- Standard care (No Intervention): Participants assigned to 'standard care' will receive the standard care required as determined by the treating team and will not be treated with nebulised heparin.

INTERVENTIONS:
Drug: Unfractionated Heparin — Heparin sodium will be administered as a nebulised aerosol dose of 25,000 IU heparin three times a day (TDS) via an Aerogen Solo (Aerogen, Ireland) vibrating mesh aerosol drug nebulizer.
  Other Names: Heparin
  Arms: Nebulised heparin

SUMMARY:
Investigator-initiated, multi-centre, randomised, open-label trial of nebulised heparin sodium in addition to standard care compared to standard care alone in hospitalised patients with COVID-19 infection.

DETAILED DESCRIPTION:
Heparin has been used as a medicine for over 75 years. It is used mostly as an anticoagulant (blood thinner), injected under the skin or infused into a vein to prevent or treat large blood clots.

Most patients who are eligible for this study are already receiving heparin administered under the skin or into a vein, and this treatment would continue after enrolment in the study, as determined by the treating doctors according to best practice.

In this study heparin is administered using a nebuliser. A nebuliser is a device that changes a fluid into a mist of tiny droplets so it can be easily breathed into the lungs. A nebuliser is a commonly used and effective way of giving medications that work in the lungs. Nebulised heparin is not currently a standard treatment, but there are good reasons to think it could help.

Lung infections, including COVID-19, cause the widespread formation of tiny blood clots in the small blood vessels and air sacs of the lungs, which make breathing difficult and lead to lung damage. Previous studies of patients with serious breathing problems due to pneumonia and other conditions found that nebulised heparin reduced the formation of small blood clots in the lungs, reduced the amount of injury to the lungs and hastened recovery with faster return to living at home. The virus that causes COVID-19 (the SARS-CoV-2 virus) has 'spikes' on its surface that enable it to attach to cells of the body and enter those cells. Another way that nebulised heparin might help is by sticking to these spikes on the virus and inhibiting the ability of the virus to enter the cells.

The main aim is to determine if nebulised heparin reduces the chance that a patient needs help with their breathing from a mechanical ventilator. Other aims are to determine if nebulised heparin increases the chances of surviving and of getting better quicker.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Currently admitted to hospital
* There is a positive sample for COVID-19 within the past 14 days. The sample can be a nasal or pharyngeal swab, sputum, tracheal aspirate, bronchoalveolar lavage, or another sample from the patient
* Requiring oxygenation according to the modified ordinal clinical scale 4-5

Exclusion Criteria:

* Intubated and on mechanical ventilation, or requiring immediate intubation as per the treating clinician's assessment
* Heparin allergy or heparin-induced thrombocytopaenia
* Activated partial thromboplastin time (APTT) > 120 seconds, not due to anticoagulant therapy and does not correct with administration of fresh frozen plasma
* Platelet count < 20 x 10^9 per L within 48 hours of randomisation
* Pulmonary bleeding or uncontrolled bleeding within 48 hours of randomisation
* Known or suspected pregnancy
* Acute brain injury that may result in long-term disability
* Myopathy, spinal cord injury, or nerve injury or disease with a likely prolonged incapacity to breathe independently e.g. Guillain-Barre syndrome
* Treatment limitations in place, i.e. not for intubation, not for ICU admission
* Death is imminent or inevitable within 24 hours
* Clinician objection
* Participant consent declined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Intubation | 28 days
  The primary outcome is intubation (or death, for patients who died before intubation) before or at day 28 after randomisation.

SECONDARY OUTCOMES:
Mortality | 60 days
  Survival to hospital discharge censored at day 60
Oxygenation | 28 days
  Daily ratio of oxygen saturation by pulse oximetry (SpO2) to the fraction of inspired oxygen (FiO2): (SpO2/FiO2 ratio, highest and lowest levels)
Length of hospitalisation | 60 days
  Duration of hospital length of stay censored at day 60

OTHER OUTCOMES:
Ventilator free days | 60 days
  The number of days without invasive mechanical ventilation censored at day 60
Length of Intensive Care Unit admission | 60 days
  Duration of intensive care unit (ICU) admission censored at day 60
Incidence of bleeding | Day 21
  The rate of bleeding including pulmonary bleeding or other major bleeding assessed daily during intervention censored at 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Frank MP van Haren, PhD, Principal Investigator — Australian National University
Locations (1):
- St George Hospital, Kogarah, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Planned international meta-trial see NCT04635241
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: real-time

REFERENCES:
- [Background] van Haren FMP, Page C, Laffey JG, Artigas A, Camprubi-Rimblas M, Nunes Q, Smith R, Shute J, Carroll M, Tree J, Carroll M, Singh D, Wilkinson T, Dixon B. Nebulised heparin as a treatment for COVID-19: scientific rationale and a call for randomised evidence. Crit Care. 2020 Jul 22;24(1):454. doi: 10.1186/s13054-020-03148-2. PMID 32698853
- [Background] van Haren FMP, Richardson A, Yoon HJ, Artigas A, Laffey JG, Dixon B, Smith R, Vilaseca AB, Barbera RA, Ismail TI, Mahrous RS, Badr M, De Nucci G, Sverdloff C, van Loon LM, Camprubi-Rimblas M, Cosgrave DW, Smoot TL, Staas S, Sann K, Sas C, Belani A, Hillman C, Shute J, Carroll M, Wilkinson T, Carroll M, Singh D, Page C. INHALEd nebulised unfractionated HEParin for the treatment of hospitalised patients with COVID-19 (INHALE-HEP): Protocol and statistical analysis plan for an investigator-initiated international metatrial of randomised studies. Br J Clin Pharmacol. 2021 Aug;87(8):3075-3091. doi: 10.1111/bcp.14714. Epub 2021 Jan 19. PMID 33377218